CLINICAL TRIAL: NCT03734679
Title: A Prospective, Multi-Center, Single-Arm Study to Assess the Safety and Performance of the Surmodics Drug Coated Balloon in the Treatment of Subjects With Obstructive Lesions of Arteriovenous Fistulae for Hemodialysis, Including Native or Synthetic Grafts
Brief Title: Safety and Efficacy of the SurVeil™ Drug-Coated Balloon (AVess FIH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SurModics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUR18-001
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Results first posted 2022-09-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Hemodialysis Access Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Surveil drug coated balloon (Experimental)
  Interventions: Device: SurVeil Drug Coated Balloon

INTERVENTIONS:
Device: SurVeil Drug Coated Balloon — Angioplasty procedure with a paclitaxel-coated, percutaneous transluminal angioplasty (PTA) balloon catheter.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the SurVeil DCB in subjects with obstructive lesions of arteriovenous fistulae for hemodialysis.

DETAILED DESCRIPTION:
AVess FIH is a prospective, multi-center, single arm, first-in-man feasibility study evaluating up to 15 subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥18 years of age.
2. Native AV fistula has been created ≥60 days prior to the index procedure.
3. AV fistula, located in the arm, has undergone one or more successful hemodialysis sessions.
4. Target de novo or non-stented restenotic lesion consisting of a ≥50% stenosis by operator visual estimate.
5. Fistula vessel diameter ≥5 mm and ≤7 mm by operator visual estimate.
6. Target lesion or tandem lesion ≤120 mm in total length by operator visual estimate.
7. Successful pre-dilatation of the target lesion. Defined as crossing of the guide wire AND pre-dilatation with a PTA balloon resulting in: residual stenosis of ≤30% and dissection ≤ Grade B
8. Subject has provided written informed consent and is willing to comply with study follow-up requirements.
9. Subject has a life expectancy of ≥1 year

Exclusion Criteria:

1. Subject has a synthetic AV graft.
2. Determined by operator to have a lesion that prevents complete inflation of an angioplasty balloon.
3. Presence of pseudoaneurysm or aneurysm requiring treatment at the lesion site.
4. Target lesion is located <30 mm from any stent.
5. Thrombosis of the access site 30 days prior to procedure.
6. Surgical revision of the access site planned within 30 days of procedure.
7. Blood coagulative disorder, sepsis, or current AV access infection (white blood count ≥12,000).
8. Known contraindication (including allergic reaction) or sensitivity to antiplatelet therapy, anticoagulation therapy or paclitaxel (mild to severe cases), that cannot be adequately managed with pre-and post-procedure medication.
9. Subjects who are taking immunosuppressive therapy or are routinely taking ≥10mg of prednisone per day.
10. Scheduled for kidney transplant or peritoneal dialysis within the next 6 months post procedure.
11. Myocardial infarction 30 days prior to procedure.
12. Stroke or TIA 90 days prior to procedure.
13. Women who are pregnant, breast-feeding or intend to become pregnant or men who intend to father children during the time of the study.
14. Subject is participating in any other investigational study that has not completed primary endpoint(s) evaluation or that clinically interferes with the endpoint from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Prince of Wales Private Hospital, Randwick, New South Wales, Australia
- Auckland City Hospital, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at two sites: site 100 - Prince of Wales Hospital, NSW Australia and site 101- Auckland City Hospital, Auckland, NZ. The first subject was enrolled at Site 100 on 5 Dec 2018, and at Site 101 on 12 Feb 2019. The last subject enrolled on 20 August 2019.
Pre-assignment Details: A total of thirteen (13) subjects were consented with the EC-approved informed consent for the trial; twelve (12) were enrolled and treated within the study and one (1) subject was a screen failure.
Groups:
- SurVeil Drug Coated Balloon: Participants were recruited at two sites: site 100 - Prince of Wales Hospital, NSW Australia and site 101- Auckland City Hospital, Auckland, NZ. The first subject was enrolled at Site 100 on 5 Dec 2018, and at Site 101 on 12 Feb 2019. The last subject enrolled on 20 August 2019.
Period: Overall Study
Arm/Group | SurVeil Drug Coated Balloon
Started | 12
Completed | 11
Not Completed | 1
Not completed — Missed Visit | 1

BASELINE CHARACTERISTICS:
Groups:
- SurVeil Drug Coated Balloon: Percutaneous transluminal angioplasty will be performed using the SurVeil™ Drug Coated Balloon (SurVeil DCB).
Arm/Group | SurVeil Drug Coated Balloon
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 7
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m²] | 30.3 (6.74)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Lesion Primary Patency at 6 Months Post Procedure
Description: Freedom from clinically-driven target lesion revascularization (CD-TLR) or access thrombosis
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil Drug Coated Balloon
Number analyzed (Participants) | 12
Participants | 11

2. Secondary Outcome: Number of Participants With Absence of All Cause Death up to 30 Days (CEC Adjudicated)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil Drug Coated Balloon
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: Number and Rate of Patients With Device and Procedure Related Adverse Events (CEC Adjudicated)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil Drug Coated Balloon
Number analyzed (Participants) | 12
Participants | 1

4. Secondary Outcome: Number of Participants With Secondary Functional Patency
Description: Secondary Patency is defined as supporting hemodialysis with a pump speed of at least 300ml/min through 6 months.
Time Frame: Through 6 months
Population: Three subjects did not have secondary functional assessed at six (6) months. One subject missed the 6-month visit. One subject underwent a kidney transplant prior to the six (6) month visit, therefore, this subject was not undergoing dialysis at this time. One subject was granted a protocol waiver by the Sponsor for trial enrollment. This subject had a mature fistula that had a treatable stenotic lesion for study entry; which has not been used for dialysis through the 6-month time period.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil Drug Coated Balloon
Number analyzed (Participants) | 9
Participants | 7

5. Secondary Outcome: Number of Participants With Subsequent Reinterventions, Such as Angioplasty, Stent, Fistula, That Are Required to Maintain Target Lesion Patency (CEC-Adjudicated)
Time Frame: 30 days and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil Drug Coated Balloon
Number analyzed (Participants) | 12
Participants
  Through 30-Day visit | 0
  Through 6-Month | 1

6. Secondary Outcome: Number of Participants With Patency of Target Lesion as Defined by Duplex Ultrasound (Reported by DUS Core Lab)
Description: Patency is defined as <50% restenosis within the target lesion.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil Drug Coated Balloon
Number analyzed (Participants) | 12
Participants | 11

7. Secondary Outcome: Number of Participants With Patency of Target Lesion as Defined by Duplex Ultrasound (Reported by DUS Core Lab)
Description: Patency is defined as <50% restenosis within the target lesion.
Time Frame: 6 months
Population: Two subjects were not included in the 6-month secondary endpoint analysis. One subject missed 6-month follow-up visit. One subject required an intervention to maintain patency during the 6-month timeframe.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil Drug Coated Balloon
Number analyzed (Participants) | 10
Participants | 2

ADVERSE EVENTS:
Time Frame: All site-reported adverse events and Serious Adverse Events (Site Reported vs. CEC Adjudicated) through 6-months, including those found to be device-related (Serious Adverse Device Effect) or procedure-related
Arm/Group | Surveil Drug Coated Balloon
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surveil Drug Coated Balloon (N=12)
Renal transplant (Surgical and medical procedures) | 1 (1)
Haematoma NOS (Vascular disorders) | 1 (1)
Physical deconditioning (General disorders) | 1 (1)
Restenosis (Injury, poisoning and procedural complications) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Heel ulcer (Vascular disorders) | 1 (1)
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Ischaemia NOS (Vascular disorders) | 1 (1)
Osteomyelitis of the foot (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surveil Drug Coated Balloon (N=12)
Pain in elbow (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth pain (Gastrointestinal disorders) | 1 (1)
Viral infection NOS (Infections and infestations) | 1 (1)
Hearing loss unilateral (Ear and labyrinth disorders) | 1 (1)
Restenosis (Injury, poisoning and procedural complications) | 3 (3)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Heel ulcer (Vascular disorders) | 1 (1)
Cerebellar lesion NOS (Nervous system disorders) | 1 (1)
Cognitive impairment (Psychiatric disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Vein rupture (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees that no publication may be made until Publication of the results of the multi-center Study or 2 years after Study Completion, whichever is the sooner. The PI must give a copy of any proposed publication to the Sponsor at least 40 days prior to public release. The sponsor may provide comments on the proposed publication, which the PI will not be bound to follow them.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT03734679/Prot_SAP_000.pdf